CLINICAL TRIAL: NCT06119841
Title: A Comparison of the Outcomes of Tonsillectomy and Expansion Sphincter Pharyngoplasty Operations in Patients With Obstructive Sleep Apnea
Brief Title: Tonsillectomy and Expansion Sphincter Pharyngoplasty Operations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Sumeyra DOLUOGLU, Principal Investigator, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDoluoglu
Record Dates: First submitted 2023-10-28; First posted 2023-11-07 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Obstructive Sleep Apnea; Osa Syndrome
Keywords: Apnea-Hypopnea Index; Expansion sphincter pharyngoplasty; Obstructive sleep apnea; Tonsillectomy; Upper airway surgery
MeSH Terms: conditions — Sleep Apnea, Obstructive; Carnevale syndrome | interventions — Tonsillectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tonsillectomy (Experimental): Tonsillectomy was performed with cold dissection including the whole tonsil and capsule, and bleeding was controlled with bipolar cauterisation.
  Interventions: Procedure: Tonsillectomy
- Expansion sphincter pharyngoplasty (Experimental): In the ESP technique, following bilateral tonsillectomy with cold dissection and bleeding control with bipolar cauterisation, the palatopharyngeus muscle was identified and a superior-based muscle flap was formed by cutting the upper two-thirds of the muscle on both sides from the lower third attachment site. By opening tunnels to the anterior plica mucosa, the dissected palatopharyngeus muscle was placed in these tunnels, and was sutured to the pterygomandibular raphe with vicryl 2-0 sutures. The mucosal cuts were closed with vicryl 3-0 sutures
  Interventions: Procedure: Expansion sphincter pharyngoplasty

INTERVENTIONS:
Procedure: Tonsillectomy — Tonsillectomy was performed with cold dissection including the whole tonsil and capsule, and bleeding was controlled with bipolar cauterisation.
  Arms: Tonsillectomy
Procedure: Expansion sphincter pharyngoplasty — In the ESP technique, following bilateral tonsillectomy with cold dissection and bleeding control with bipolar cauterisation, the palatopharyngeus muscle was identified and a superior-based muscle flap was formed by cutting the upper two-thirds of the muscle on both sides from the lower third attachment site. By opening tunnels to the anterior plica mucosa, the dissected palatopharyngeus muscle was placed in these tunnels, and was sutured to the pterygomandibular raphe with vicryl 2-0 sutures. The mucosal cuts were closed with vicryl 3-0 sutures
  Arms: Expansion sphincter pharyngoplasty

SUMMARY:
Background: To compare the efficacy of tonsillectomy and expansion sphincter pharyngoplasty (ESP) in the surgical treatment of obstructive sleep apnea (OSA).

Methods: Patients with Friedman grade III-IV tonsil hypertrophy and OSA diagnosed with polysomnography were separated into two groups according to the surgery performed, as the classic tonsillectomy group (Group 1) and the ESP group (Group 2). The primary endpoint of the study was to determine the Apnea-Hypopnea Index (AHI) value. The preoperative and postoperative AHI scores and the decreases in these scores were noted. The change in AHI was calculated as a percentage (preoperative AHI - postoperative AHI/ preoperative AHI x 100) and the two groups were compared. An AHI value of <10 events/hour was accepted as cure.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a frequently seen sleep disorder characterised by the stopping or decrease of air flow, which occurs with the collapse of the upper airway during sleep. The upper airway can be described as an empty tube and if the air passing through this tube decreases or stops, an increase in negative pressure occurs, especially in the soft palate and lateral pharyngeal wall, causing pharyngeal collapse The increase in airway resistance because of both the upper airway collapse and increase in negative pressure can be a reason for loud snoring and apnea, and if not treated can also cause systemic complications. Upper airway obstruction formed in OSA can be due to structural anatomic factors or to abnormal upper airway motor tonus. The obstruction in the upper airway can occur in a single or several anatomic regions such as the soft palate, uvula, palatine tonsils, or tongue root. Treatment modalities include lifestyle changes, continuous positive airway pressure (CPAP), surgery, and intra-oral devices. The main aim of all treatments is to expand the upper airway and attempt to reduce airway collapse. In the surgical treatment applied for this purpose, it is aimed to remove pharyngeal tissue that narrows the upper airway, increase the stability of the pharyngeal air column, and expand the pharyngeal lumen.

The lateral pharyngeal wall has a complex structure including several pharyngeal muscles such as the palatopharyngeus, superior pharyngeal constrictor, and palatoglossus, and lymphoid tissue, and the palatine tonsils. In a previous study, the clinical importance was stated of lateral pharyngeal wall collapse in the pathogenesis of OSA. It was suggested in that study that the lateral pharyngeal wall could collapse more easily especially in patients with severe OSA compared to those without or with mild OSA, and because of this collapse, the narrowed lateral pharyngeal wall could be an independent risk factor affecting OSA. The palatine tonsils, especially those of Friedman grade III-IV dimensions, which occupy a large space in the lateral pharyngeal wall, seem to be a factor causing collapse. In OSA patients with grade III-IV tonsil hypertrophy, classic tonsillectomy is recommended as first-line treatment and is still the gold standard surgical method. However, sometimes tonsillectomy remains insufficient in the treatment of OSA. Therefore, to be able to prevent lateral pharyngeal wall collapse and increase stability, surgical techniques have been investigated, and lateral pharyngoplasty, relocation pharyngoplasty, and most recently, expansion sphincter pharyngoplasty (ESP) have been defined. A previous study has reported that ESP is a suitable surgical procedure for patients with moderate or severe OSA who have severe palatal circumferential narrowing and greater lateral pharyngeal wall thickness. A meta-analysis that included 5 studies also emphasized that ESP was an effective surgical treatment for OSA patients. However, to the best of our knowledge, there is no study in the literature that has shown whether or not this surgical technique is superior to classical tonsillectomy. The need for this method, which is more major surgery than classic tonsillectomy, is not clear. Therefore, the aim of this study was to investigate and compare the surgical success of classic tonsillectomy and ESP in OSA surgery performed on a patient series in our hospital.

The study was conducted in the Ear, Nose, and Throat (ENT) Clinic of a city hospital. A full ENT examination was made of patients with suspected OSA who presented with complaints of loud snoring, witnessed apnea, and daytime sleepiness. The obstruction localisation was evaluated using the Müller manoeuvre during the endoscopic examination and only patients with lateral pharyngeal collapse were included in the study.Then preoperative polysomnography (PSG) was performed on the patients with Friedman grade III-IV tonsil hypertrophy. The study included patients aged >18 years with an Apnea-Hypopnea Index (AHI) value of ≥10. Patients were excluded from the study if they had not undergone preoperative or postoperative PSG, if they had a craniofacial anomaly such as evident retrognathia, any severe cardiac, respiratory, or neurological disease, or were determined with an evident obstruction at the tongue base level in the endoscopic examination.

The patients who underwent surgery for a diagnosis of OSA were separated into two groups as the classic tonsillectomy (Group 1) and ESP (Group 2) groups. All the operations were performed by two surgeons experienced in this subject (MM-AI). The patients were hospitalised for at least 2 days postoperatively, with hydration and pain relief provided.

The primary endpoint of the study was defined as the AHI score. The patients were separated into 3 subgroups according to the severity of OSA determined in the PSG recording: mild (AHI ≥ 10 and <15 events/hr), moderate (AHI ≥15 and <30 events/hr), and severe (AHI ≥ 30 events/hr). The preoperative and postoperative AHI scores and the decreases in these scores were noted. The change in AHI was calculated as a percentage (preoperative AHI - postoperative AHI/ preoperative AHI x 100) and the two groups were compared. An AHI value of <10 events/hr was accepted as cure. Success was considered as postoperative AHI <20 events/hr or a 50% reduction in the preoperative AHI.

The daytime sleepiness status of the patients was evaluated using the Epworth Sleepiness Scale (ESS). A record was made for each patient of body mass index (BMI), smoking status and alcohol consumption, and history of comorbidities. At postoperative 6 months, PSG was repeated, the ESS was applied, and BMI was recorded.

All the operations were performed under general anaesthesia. Tonsillectomy was performed with cold dissection including the whole tonsil and capsule, and bleeding was controlled with bipolar cauterisation. In the ESP technique, following bilateral tonsillectomy with cold dissection and bleeding control with bipolar cauterisation, the palatopharyngeus muscle was identified and a superior-based muscle flap was formed by cutting the upper two-thirds of the muscle on both sides from the lower third attachment site. By opening tunnels to the anterior plica mucosa, the dissected palatopharyngeus muscle was placed in these tunnels, and was sutured to the pterygomandibular raphe with vicryl 2-0 sutures. The mucosal cuts were closed with vicryl 3-0 sutures. All the patients were discharged on postoperative day 2. Follow-up examinations were made at the end of postoperative 1 week, 1, 3, and 6 months. The Clavien-Dindo system was used to evaluate complications.

Statistical Analysis Data analysis was performed using SPSS for Windows, version 26 software (SPSS Inc., Chicago, IL, USA). Continuous variables were reported as median (minimum-maximum) values, and categorical variables as number (n) and percentage (%). Nominal variables were assessed using the Pearson's Chi-square or Fisher's exact test. For parameters that did not show normal distribution, the Mann-Whitney U test was applied in comparisons. The Wilcoxon signed-rank test was used to compare pre- and post-surgery AHI scores. A value of p< 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* patients aged >27 years
* Apnea-Hypopnea Index (AHI) value of ≥10.

Exclusion Criteria:

* absent preoperative and/or postoperative PSG
* craniofacial anomaly such as evident retrognathia
* severe cardiac, respiratory, or neurological disease
* an evident obstruction at the tongue base level in the endoscopic examination

Ages: 27 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index (AHI) | 1 hour
  The patients were separated into 3 subgroups according to the severity of OSA determined in the PSG recording: mild (AHI ≥ 10 and <15 events/hr), moderate (AHI ≥15 and <30 events/hr), and severe (AHI ≥ 30 events/hr). The preoperative and postoperative AHI scores and the decreases in these scores were noted. The change in AHI was calculated as a percentage (preoperative AHI - postoperative AHI/ preoperative AHI x 100) and the two groups were compared. An AHI value of <10 events/hr was accepted as cure. Success was considered as postoperative AHI <20 events/hr or a 50% reduction in the preoperative AHI.

CONTACTS AND LOCATIONS:
Overall Officials: Gokhan Toptas, MD, Study Chair — Saglik Bilimleri Universitesi
Locations (1):
- Ankara Etlik City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
To compare the efficacy of tonsillectomy and expansion sphincter pharyngoplasty (ESP) in the surgical treatment of obstructive sleep apnea (OSA).